CLINICAL TRIAL: NCT05283941
Title: Pistachios and Neural Macular Pigment; a Randomized Controlled Trial
Brief Title: Pistachios and Neural Macular Pigment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tufts University (Other)
Collaborators: American Pistachio Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N322001 FSU054
Record Dates: First submitted 2022-02-22; First posted 2022-03-17 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases
Keywords: age related macular degeneration; lutein; zeaxanthin; pistachios; macular pigment; AMD
MeSH Terms: conditions — Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pistachio Group (Experimental): The pistachio group will receive pistachio nuts in 2-ounce packs. This group will consume one pack every day over the course of the 12-week study.
  Interventions: Dietary Supplement: Pistachio Group
- Control (Usual Diet) Group (No Intervention): The control group will not receive pistachio nuts. They will be asked to make no changes and continue to eat their regular diet.

INTERVENTIONS:
Dietary Supplement: Pistachio Group — Consumption of 2-ounce packs of pistachio nuts, daily, for 12 weeks.
  Arms: Pistachio Group

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of irreversible vision loss as people age. Studies have shown that lutein and zeaxanthin, nutrients found in green leafy vegetables and egg yolks, can help protect against AMD in older adults. These nutrients form a pigment in the retina (macular pigment) that can help protect the retina from light damage. Pistachios are rich sources of both lutein and zeaxanthin; thus, dietary intake of pistachios could serve as a beneficial food source for eye health.

DETAILED DESCRIPTION:
Lutein and its isomer zeaxanthin (L/Z) are dietary carotenoids that cross the blood brain barrier and exclusively accumulate in the macular region of the retina, where they are referred to as macular pigment (MP). MP density (MPD) has been reported to be significantly related to decreased risk of age-related macular degeneration as well as cognitive function in both young and older adults. Studies in non-human primates and humans find that MPD is significantly related to lutein brain concentrations. MPD, a non-invasive measure, is thus a biomarker for brain concentrations of L/Z. This may be of interest given the report that L/Z concentrations in the older adult brain are positively related to a variety of pre mortem cognitive measures. Furthermore, L/Z supplementation was found to significantly improve verbal fluency scores in healthy older adults. Pistachios are a bioavailable source of L/Z. L/Z are transported in the circulation primarily on high density lipoproteins (HDL) and HDL levels were found to be significantly related to MPD. Thus, increasing dietary intake of L/Z as well as changing lipoprotein levels may impact MPD. This is of interest given that a pistachio enriched diet has been reported to improve lipid profile in healthy and mild hypercholesterolemic patients. Based on the sum of these findings, the objective of this study was to investigate the effect of a long-term pistachio intervention on MPD.

The overall goal of the proposal is to determine whether the consumption of pistachios is a practical way to increase L/Z status. This will primarily be accomplished by performing a nutritional study to demonstrate that pistachios are a bioavailable source of L/Z to neural tissue (i.e., MP). Cross-sectional and intervention studies report a significant relationship between L/Z levels and ocular and cognitive health. Current L/Z intakes in the U.S. are lower than levels associated with health. This randomized, parallel study will test the efficacy of pistachios on increasing L/Z neural status (i.e., MPD).

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women, aged 40 - 70 years
2. Body Mass Index (BMI): 20.0 - 36.9 kg/m2
3. Low macular pigment density at baseline (<0.5 OD)
4. Low lutein and zeaxanthin intake at baseline (<2 mg/d)

Exclusion Criteria:

1. Inability to perform the heteroflicker photometry procedures with or without corrective lenses (i.e. glasses or contact lenses) during in-house screening.
2. History of (self-reported):

   * Fat malabsorption
   * Use of drugs that interfere with fat absorption or metabolism
   * Tree nut allergy
   * Eye disease, including macular degeneration and cataracts
   * Small bowel disease or resection
   * Atrophic gastritis
   * Hyperlipidemia
   * Insulin-requiring diabetes
   * > 14 alcoholic drinks per week
   * Pancreatic disease
   * Bleeding disorders
   * Pregnancy (or hoping to become pregnant during participation in the study)
   * Carotenoid or fatty acid dietary supplements within 2 months of the study
   * Non-English speaker
   * Any condition that would make it unlikely that the participant would be able to complete the requirements of the study.

Individuals on lipid-lowering medication will be considered if they maintain their regimen throughout the study and meet all inclusion/exclusion criteria.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Macular Pigment (MP) Density over 12 weeks | Measured at baseline, 6 weeks and 12 weeks.
  A non-invasive psychophysical technique, known as heterochromatic flicker photometry (HFP), will be used to measure MP density of the retina.

SECONDARY OUTCOMES:
Serum concentrations of lutein and zeaxanthin (dietary carotenoids) | Measured at baseline and 12 weeks.
  Serum carotenoids will be measured by HPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Scott, Principal Investigator — Tufts University
Locations (1):
- Clinical and Translational Research Center (CTRC) - Tufts, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scott TM, Ogunbodede O, McKay DL, Johnson EJ. Pistachio Consumption Increases Macular Pigment Optical Density in Healthy Adults: A Randomized Controlled Trial. J Nutr. 2025 Jan;155(1):168-174. doi: 10.1016/j.tjnut.2024.10.022. Epub 2024 Oct 18. PMID 39426460